CLINICAL TRIAL: NCT05957562
Title: Azygos Vein Preservation Revisited: Impact on Early Outcomes After Repair of Esophageal Atresia/ Tracheo-Esophageal Fistula in Newborns: A Randomized Controlled Study
Brief Title: Azygos Vein Preservation; Its Impact on Early Outcomes After Neonatal EA/TOF Repair
Acronym: EArAzygousvp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dr. Muhammad Abdelhafez Mahmoud, MD (Other)
Responsible Party: Sponsor-Investigator, dr. Muhammad Abdelhafez Mahmoud, MD, Lecturer of pediatric surgery, Al-Azhar Faculty of Medicine, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AlAzharEArepairAzygouspreserve
Record Dates: First submitted 2023-07-09; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Azygos Vein Preservation Versus Disconnection; Tracheo-Esophageal Fistula With Atresia of Esophagus; Leak, Anastomotic; Stricture Esophagus; Pneumonitis; Postoperative
Keywords: Esophageal Atresia,; Tracheoesophageal fistula,; Preservation of the Azygos vein,; Division of Azygos vein,; Pediatrics
MeSH Terms: conditions — Esophageal atresia with or without tracheoesophageal fistula; Anastomotic Leak; Esophageal Stenosis; Pneumonia; Esophageal Atresia; Tracheoesophageal Fistula

STUDY DESIGN:
Intervention Model Description: This randomized controlled study conducted to assess the technical feasibility and surgical outcomes of one stage surgical repair, either with Azygos vein preservation or with Azygous vein disconnection, in newborns diagnosed with Esophageal Atresia and tracheoesophageal fistula. It includes 64 neonates with TOF/EA who will be randomly divided (using the sealed closed envelope method) into two equal groups, each group will include 34 neonatal patients
Who Masked: Participant
Masking Description: single (participants will choose from sealed closed envelopes)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EA/TOF primary repair with Azygos vein preservation (Active Comparator): primary esophagoesophagostomy with azygous vein preservation technique and will be done for 32 neonates with EA/TOF amenable for primary repair
  Interventions: Procedure: EA/TOF primary repair with Azygos vein preservation
- EA/TOF primary repair with Azygos vein sacrifice (disconnection) (Active Comparator): primary esophagoesophagostomy with azygous vein disconnection ordinary technique and will be done for 32 neonates with EA/TOF suitable for primary repair
  Interventions: Procedure: EA/TOF primary repair with Azygos vein sacrifice (disconnection)

INTERVENTIONS:
Procedure: EA/TOF primary repair with Azygos vein preservation — primary repair of EA/TOF with either azygous vein preservation or disconnection (to assess the effects and expected benefits of the former technique on viability of the repair and decrease of postoperative early complications and mortality rate)
  Arms: EA/TOF primary repair with Azygos vein preservation
Procedure: EA/TOF primary repair with Azygos vein sacrifice (disconnection) — primary repair of EA/TOF with either azygous vein preservation or disconnection (to assess the effects and expected benefits of the former technique on viability of the repair and decrease of postoperative early complications and mortality rate)
  Arms: EA/TOF primary repair with Azygos vein sacrifice (disconnection)

SUMMARY:
Azygos vein preservation revisited: impact on early outcomes after repair of Esophageal atresia/ Tracheo-Esophageal Fistula in newborns. A randomized controlled study.

DETAILED DESCRIPTION:
Since the first successful repair of esophageal atresia/tracheoesophageal fistula was performed approximately eight decades ago, surgeons have made considerable technical advances in solving intraoperative surgical challenges and reducing postoperative complications. According to some surgeons, the advantage of maintaining the Azygos vein makes this modification attractive. This study aimed to explore the benefits of retaining the Azygos vein during surgery for Esophageal Atresia with tracheoesophageal fistula, to emphasize its advantages in terms of reducing anastomotic leak, stricture, and other postoperative outcomes.

Patients and Methods: This prospective randomized study was conducted between April 2020 and April 2023. The study included all newborns with (EA & TEF) eligible for primary repair, patients were randomly assigned to either Group A or Group B. (Group A) patients who underwent Azygos vein preservation during TEF repair, whereas the remaining patients (Group B) had Azygos vein disconnection.

Statistical analysis: The Statistical Package for Social Sciences (SPSS) (version 23.0, IBM Corp IBM Corp., Armonk, NY, USA) was used for statistical analysis. The chi-square test (X2) was used to compare qualitative data in the groups, while an independent-sample t-test was used to compare quantitative data between groups. The degree of confidence was set at 95%. The p-value was considered significant at a level of 0.05.

Discussion: will focus on advantages of azygous vein preservation on intactness of esophageal anastomosis, retaining the venous drainage of the bronchial system, and chest wall. Points of discussion will include effects of Azygous vein preservation on incidence of postoperative pneumonitis, anastomotic leakage and stricture rate, and mortality rate. The results obtained from this study will be compared between both groups and with those reported in the literature.

Finally, the investigators will conclude the reconstructive technique that gives the better results and least morbidity.

ELIGIBILITY:
Inclusion Criteria:

* all neonates suitable for primary repair of Esophageal Atresia and tracheoesophageal fistula

Exclusion Criteria:

* long gap esophageal atresia (> 3 cm)
* esophageal atresia without tracheoesophageal fistula

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
gap between the pouches after mobilization | 2 years
  missed distance between the mobilized esophageal pouches in centimeters
operative time | 2 years
  operative time in minutes
early postoperative pneumonia | 35 months
  postoperative pneumonitis in number
early postoperative anastomotic leak | 35 months
  anastomotic leakage rate in number
early postoperative anastomotic stricture | 35 months
  anastomotic stricture rate in number
mortality | 35 months
  mortality rate in number

SECONDARY OUTCOMES:
gestational age | 2 years
  gestational age in weeks
sex | 2 years
  patient's gender in number
associated congenital anomalies | 2 years
  associated congenital anomalies in number
associated anomalies | 2 years
  associated congenital anomalies in percentage of cases

OTHER OUTCOMES:
Spitz classification | 2 years
  Spitz classification of mortality risk of TOF/EA in number

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshamy, MD, Study Chair — Pediatric Surgery Unit-Department of Surgery, Al-Azhar University, Assuit, Egypt
Locations (1):
- Pediatric Surgery Department, Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analyzed during the current study are available from the corresponding author but could not be sent owing to the medicolegal aspect of the hospital policy.

REFERENCES:
- Available data/document: Study Protocol: orcid.org/0000-0003-0558-6402 — http://orcid.org/0000-0003-0558-6402